CLINICAL TRIAL: NCT05103605
Title: Positioning, Utilization and Effectiveness of Osimertinib in First Line in Real-life Therapeutic Strategy in France Prospective Cohort of Locally Advanced and Metastatic Non-Small Cell Lung Cancer Patients With Activating EGFR Mutations
Brief Title: Prospective Cohort of Locally Advanced and Metastatic Non-Small Cell Lung Cancer Patients With Activating EGFR Mutations
Acronym: POSITHES
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00017
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

INTERVENTIONS:
Drug: Osimertinib — Single arm treated by osimertinib
  Other Names: TAGRISSO

SUMMARY:
This is an observational multicenter study. A cross-sectional descriptive study of patients with locally advanced or metastatic Non Small Cell Lung Cancer with activating EGFR mutation treated by any first line therapy will be used to identify cohort with a prospective follow-up of patients initiating a treatment by osimertinib in first line

* A cross-sectional descriptive study of all patients with locally advanced or metastatic NSCLC with activating EGFR mutation treated by any first line therapy will be collected at the study participating sites. The study which is transversal will allow to characterize the population of patients with locally advanced or metastatic NSCLC with activating EGFR mutation treated in first line, the day of first line initiation.
* Additionally, a prospective study targeting a cohort of patients focusing on patients with locally advanced or metastatic NSCLC with activating EGFR mutation initiating a treatment by osimertinib in first line will be conducted to address describe in real life conditions the 36-months overall survival, patients baseline characteristics, disease evolution, sequencing and treatment patterns, and quality of life

DETAILED DESCRIPTION:
This is an observational multicenter study combining a descriptive cross-sectional survey and a prospective cohort design to address the study objectives.

Part A is a prospective study targeting a cohort of patients focusing on patients with locally advanced or metastatic NSCLC with activating EGFR mutation initiating a treatment by osimertinib in first line will be conducted to address the primary objective of this study and remaining secondary objectives.

Part B is an additional descriptive cross-sectional survey of all patients with locally advanced or metastatic NSCLC with activating EGFR mutation treated by any first line therapy will be collected at the study participating sites. The study part which is cross sectional will allow to characterize the population of patients with locally advanced or metastatic NSCLC with activating EGFR mutation treated in first line, the day of first line initiation.

Both studies will be initiated at the same time (depending on osimertinib reimbursement in France - expected on October 2020). Part A will have an enrolment period of approximately 18 months and a follow-up period of 36 months. Part B will have an enrolment period of 12 months.

For Part A, patients must be newly treated in first line and the index date will be the day of first line treatment initiation. Patients will be followed-up for all routine visits recorded until time to second progression. After the relapse of second line therapy, patients will be followed-up every 6 months for overall survival only until 36 months.

For Part B, patients newly diagnosed with locally advanced or metastatic NSCLC who are treatment naive or patients who were diagnosed at an earlier stage but have progressed to metastatic NSCLC during the selection period will be included.

Patients will be followed up from enrolment in part A until death, loss to follow-up, withdrawal of consent or study end date, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Descriptive cross-sectional survey (Population B)

  * Adult patients (≥ 18 years old),
  * Patients newly treated in first line (1L) for locally advanced or metastatic NSCLC,
  * Patients with activating EGFR mutation-positive,
  * Patient informed and not opposed to these data collection.
* Prospective cohort (Population A)

  * Patient meeting part B inclusion criteria,
  * Patients newly treated in 1L by osimertinib,
  * Patient with common EGFR mutation-positive (exon 19 deletion or L858R mutation, alone or co-occuring with other EGFR mutations).

Exclusion Criteria (Population A):

* Patients enrolled in interventional clinical trials (first line treatment for a NSCLC) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study combining a descriptive cross-sectional survey (part B) and a prospective cohort design (part A).
  Patients with locally advanced or metastatic Non Small Cell Lung Cancer (NSCLC) with activating EGFR mutation initiating a treatment by osimertinib in first line (Population A)
  Patients with locally advanced or metastatic NSCLC with activating EGFR mutation treated by any first line therapy (population B)
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 36 months
  36-months overall survival defined as time from index date until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Auliac, Principal Investigator — CHI Creteil, France
Locations (46):
- France (46):
  - Research Site, Abbeville
  - Research Site, Aix-en-Provence
  - Research Site, Angers
  - Research Site, Antibes
  - Research Site, Avignon
  - Research Site, Bastia
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Brest
  - Research Site, Cannes
  - Research Site, Chambéry
  - Research Site, Chauny
  - Research Site, Cholet
  - Research Site, Clermont-Ferrand
  - Research Site, Colmar
  - Research Site, Contamine-sur-Arve
  - Research Site, Créteil
  - Research Site, Elbeuf
  - Research Site, Epagny METZ Tessy
  - Research Site, Évreux
  - Research Site, La Roche-sur-Yon
  - Research Site, Libourne
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Meaux
  - Research Site, Mulhouse
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Quimper
  - Research Site, Reims
  - Research Site, Rouen
  - Research Site, Saint-Denis
  - Research Site, Saint-Grégoire
  - Research Site, Saint-Pierre
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Valenciennes
  - Research Site, Vannes
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villenave-dornon
  - Research Site, Villeurbanne

IPD SHARING:
Plan to Share IPD: No